CLINICAL TRIAL: NCT06582147
Title: Implementing a Social Determinants of Health Screening and Referral Care Model in the Neonatal Intensive Care Unit
Brief Title: The Social Determinants of Health Screening and Referral Project
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Margaret Parker, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000543; 5R01HD104772 (NIH)
Record Dates: First submitted 2024-08-14; First posted 2024-09-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Preterm Birth
Keywords: Neonatal intensive care unit (NICU); Social determinants of health (SDOH); WE CARE; SDoH screening and referral; Mother-infant dyads; Maternal depression; Safety net hospitals
MeSH Terms: conditions — Premature Birth | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Hybrid effectiveness- implementation stepped wedge cluster randomized trial (SW-CRT) using the Proctor Conceptual Model of Implementation Research.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social needs screening and referral care (Other): As a step wedge cluster randomized trial all sites will be assigned to receive the intervention in a randomized order. There is no difference in the intervention by site, the only difference is the timing of the beginning of the intervention. Therefore, we have only identified one arm.
  Interventions: Other: Implementation of social determinants of health screening and referral

INTERVENTIONS:
Other: Implementation of social determinants of health screening and referral — WE CARE is a relatively simple, low-intensity intervention that has two key components: (1) screening individuals using the WE CARE SDOH Screener for unmet social needs, and (2) providing individuals who have unmet social needs with SDOH Community Resource sheets
  Other Names: WE CARE

SUMMARY:
Up to a quarter of the families with preterm infants have unmet social needs, such as housing or job insecurity, which represent adverse social determinants of health (SDOH). Preterm infants are especially vulnerable to the social conditions they grow up in, with sustained impacts on function across multiple organ systems. The goal of this study is to translate an established model of SDOH screening and referral from the outpatient setting to the NICU, thereby maximizing the potential to offset the effects of adverse SDOH on vulnerable mother-preterm infant dyads.

DETAILED DESCRIPTION:
The goal of this study is to implement SDOH screening and referral models in 7 safety net NICUs, examining their potential to offset the effects of adverse SDOH for a highly vulnerable population at the earliest stages of life. The investigators propose a hybrid effectiveness-implementation stepped wedge cluster randomized trial using the Proctor Conceptual Model of Implementation Research. The investigators will follow a cohort of 882 mother-infant dyads longitudinally for 12 months after NICU discharge to examine family, maternal, and infant outcomes. Each site will participate in three phases: usual, experimental, and sustainment.

The study aims are to:

Aim 1: Examine the implementation of SDOH screening and referral models into the NICU (acceptability, feasibility, penetration, equity, and sustainability).

Aim 2: Examine the effectiveness and equity of SDOH screening and referral models in the NICU setting on parental receipt of community resources for unmet social needs 3 months post-NICU discharge.

Aim 3: Explore the effectiveness of SDOH screening and referral models in the NICU to improve (a) maternal mental health (depression) and (b) health and developmental outcomes of preterm infants (quality of life, growth, development, and respiratory disease) during the 12 months post-NICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Infant gestational age <34 weeks' gestation; singleton or multiple.
* Infant hospitalized for at least 14 days of life (to allow for SDOH screening/referral and contact with resources if applicable).
* Mother and infant are alive.
* Mother speaks and reads English or Spanish.
* Infant will be discharged home from the NICU (to allow for follow-up).
* Mother will care for her infant(s) at home in the US for at least 12 months after discharge from the NICU.

Exclusion Criteria:

* Mothers or infants who die before anticipated infant discharge.
* Infant discharged after 52 weeks postmenstrual age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Penetration of SDOH intervention | Monthly for approximately 12 months
  Penetration is the rate of administration of social needs screener and appropriate referral for community resources to eligible families.
Receipt of ANY Community Resource | 3 months Post-NICU discharge
  Receipt of any community resource as collected via participant survey specifying receipt of the resource.

SECONDARY OUTCOMES:
Acceptability of SDOH intervention | Approximately 7, 9, and 12 months
  Mean score on Acceptability of Intervention Measure (AIM), which is a 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). The score is calculated mean, and higher scores are associated with better acceptability. (Minimum score is 4, maximum score is 20).
Feasibility of SDOH intervention | Approximately 7, 9, and 12 months.
  Mean score on Feasibility of Intervention Measure (FIM) is A 4-item instrument to assess perceived intervention feasibility. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean, and higher scores are associated with better feasibility. (Minimum score is 4, maximum score is 20).
Sustainability of SDOH intervention | Monthly for approximately 6 months.
  Number of individuals who continued to get screened after active intervention is complete.
Equity of implementation | Monthly for approximately 18 months (during both penetration and sustainability).
  Penetration rate by maternal demographics.
Equity of receipt of community resources | 3 months Post-NICU discharge
  Rate of receipt of community resources by maternal demographics
SDOH Risk | Baseline, 3 months, 6 months, and 12 months Post-NICU discharge
  Any social need or change in social need for housing, food, utilities, childcare, employment, transportation, or education was collected via participant survey.
SDOH Desire Assistance | Baseline, 3 months, 6 months, and 12 months Post-NICU discharge
  Any desired assistance or change in desired assistance for housing, food, utilities, childcare, employment, transportation, and education was collected via participant survey.
SDOH Community Resource | Baseline, 3 months, 6 months, and 12 months Post-NICU discharge
  Number of individuals who received any community resource (housing, food, utilities, education, employment, childcare, transportation).
Family Economic Pressure | Baseline, 3 months, 6 months, and 12 months Post-NICU discharge
  The Family Economic Pressure scale is a 2-item measure that is scored and summed together. Scores on Measures A and B are from the Economic Pressure Scale. Higher levels indicate higher economic hardship. (Minimum score is 6, maximum score is 30).
Maternal Wellbeing | Baseline, 3 months, 6 months, and 12 months Post-NICU discharge
  Rating of current overall health
Postpartum maternal primary care utilization | 3 months, 6 months, and 12 months Post-NICU discharge
  Number of appointments with a primary care provider
Maternal Postpartum Obstetric Care Utilization | 3 months, 6 months, and 12 months Post-NICU discharge
  Number of appointments with a maternal postpartum obstetric provider
Maternal emergency room utilization | 3 months, 6 months, and 12 months Post-NICU discharge
  Number of emergency room visits.
Maternal hospital readmission | 3 months, 6 months, and 12 months Post-NICU discharge
  Number of overnight hospital readmissions
Maternal Depression | Baseline, 3 months, 6 months, and 12 months Post-NICU discharge
  Overall score on Personal Health Questionnaire Depression Scale (PHQ8), an 8-item instrument with 4 category Likert scale responses from 0 to 4 where 0=not at all and 4=daily. Scores can range from 0 to 32. Higher scores are associated with greater levels of maternal depression.
Length of Lactation | Baseline, 3 months, 6 months, and 12 months Post-NICU discharge
  Duration of milk production in months
Infant primary care utilization | 3 months, 6 months, and 12 months Post-NICU discharge
  Number of appointments with a primary care provider
Infant utilization of emergency care | 3 months, 6 months, and 12 months Post-NICU discharge
  Number of emergency room visits
Infant hospital readmission | 3 months, 6 months, and 12 months Post-NICU discharge
  Number of overnight hospital readmissions
Receipt of necessary infant services and equipment | 3 months, 6 months, and 12 months Post-NICU discharge
  The proportion of individuals who receive services and equipment among those individuals who indicate needing services and equipment on the national survey of children with special healthcare needs
Infant Respiratory Symptoms (shortness of breath, wheezing, coughing, clinically demonstrated need for oral corticosteroids) | 3 months, 6 months, and 12 months Post-NICU discharge
  Overall score on Test for Respiratory and Asthma Control in Kids. Each item is scored from 0 to 20 points on a 5-point Likert-type scale for a total score ranging from 0 to 100. Higher scores indicate better respiratory control.
Infant growth | Baseline, 3 months, 6 months, and 12 months Post-NICU discharge
  Weight for age z-score change
Infant Quality of Life | 3 months, 6 months, and 12 months Post-NICU discharge
  Overall score on the Infant Toddler Quality of Life Questionnaire™ (ITQOL) is a 47-item short form that is scored on a scale from 0 (worst health) to 100 (best health). Higher scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Parker, MD, MPH, Principal Investigator — University of Massachusetts Chan Medical School; Mari-Lynn Drainoni, PhD, MEd, Principal Investigator — Boston University Chobanian and Avedisian School of Medicine; Arvin Garg, MD, MPH, Principal Investigator — University of Massachusetts Chan Medical School
Locations (7):
- United States (7):
  - Denver Health Hospital Authority, Denver, Colorado
  - Shands Jacksonville Medical Center, Inc. DBA UF Health Jacksonville, Jacksonville, Florida
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be submitted to the MPIs after study completion.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted to the MPIs 6 months after study completion.
Access Criteria: Access to data can be requested by qualified researchers engaging in independent scientific research. Requests must include review and approval of the research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Statement (DSA).